CLINICAL TRIAL: NCT01602848
Title: A Patient Centered Intervention to Improve Health and Reduce Medicaid Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-08-243-05-G
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: High-risk, High-cost Medicaid Services Users
Keywords: Medicaid; frequent users; heavy users; high risk; high cost; intervention to improve care and reduce Medicaid expenditures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention enrollee (Experimental): HIgh risk fee for service Medicaid recipients identified as eligible by the New York State Dept of Health and enrolled in the intensive care management and coordination intervention
  Interventions: Other: Intensive care management and coordination
- Eligible, not enrolled (No Intervention): Medicaid fee-for-service patients who are identified as eligible for the intervention but are not enrolled. These patients receive usual services provided by Medicaid.

INTERVENTIONS:
Other: Intensive care management and coordination — Care Management Teams comprised of social workers, community based care managers, and dedicated clinicians work to meet patients' needs in both the health care setting and the community. The CIDP model incorporates motivational interviewing, harm reduction, access to housing through our community partners utilizing a Housing First approach, and provides cellular phones for patients when needed, to better enable regular communication with program staff.
  Arms: Intervention enrollee

SUMMARY:
Medicaid-insured patients with frequent hospitalizations account for a disproportionate share of visits and costs, and have caught the attention of policy makers, creating an impetus for hospitals and health care providers to better understand and control associated expenditures. Many such patients have specific unmet health and social needs. Based on our extensive pilot work with this population, the New York State Department of Health recently awarded the New York City Health and Hospitals Corporation one of seven statewide contracts to implement a Chronic Illness Demonstration Project, aimed at improving care and reducing healthcare expenditures for high cost Medicaid patients. Within this framework, the investigators propose a group-randomized trial design to test whether specific outcomes related to health, functional status, and quality of life resulting from a patient-centered, intensive care coordination and management intervention correlate with improved linkage to primary care while reducing hospitalizations and emergency department visits. The investigators will then relate these benefits to program costs using standard cost-effectiveness analysis techniques. Given that there are few examples of successful interventions for this population and currently unparalleled Medicaid spending, there is an urgent need to demonstrate that interventions to improve care coordination and optimize patients' use of the health and social care system result in more efficient and less costly care.

DETAILED DESCRIPTION:
Though patients with frequent hospital admissions comprise a small percentage of all patients, they account for a disproportionate share of visits and costs. Their substantial use of health care resources is often a result of the simultaneous presence of severe medical and social co-morbidities. These high cost cases have caught the attention of policy makers, and have created a movement by states to shift Medicaid patients from fee-for-service into managed care models or "high risk" case management programs. Such state initiatives create an impetus for hospitals and health care providers to better understand and control expenditures for the highest users of health services.

The work proposed for this application will address this gap in the literature through the use of a group-randomized trial design using quantitative to evaluate outcomes. This proposal is a logical extension of our previous work: for the past three years, we have been conducting research on improving care coordination for this patient population via in-depth needs assessment, model program development, and implementation of a pilot initiative at a safety net hospital for a limited number of patients to determine feasibility. Most recently, the New York City Health and Hospitals Corporation (HHC) was awarded one of seven New York State Department of Health Chronic Illness Demonstration Project (CIDP) grants of over $5 million and spanning 3 years, to expand this work to enroll and intervene with similar high-risk patients throughout the system.

In order to evaluate the impact of the CIDP initiative, the intervention is currently designed as a group-randomized trial that will track and compare the health care utilization and costs in intervention and control groups using Medicaid claims data. However, no provision has been made for contacting or characterizing control group members, or for surveying control group members regarding issues such as depression, social support, behavioral health needs, or satisfaction with current care, leaving the question of which intervention components correlate with changes in health services utilization unanswered. The ability of the evaluation to analyze the effect of important factors we anticipate will be improved by this innovative care redesign initiative (e.g., social support, housing status) on health services utilization is thus sharply curtailed, limiting the outcomes being studied to those derivable from administrative claims data.

We thus propose to conduct an in-depth evaluation of the HHC CIDP enrollees to determine whether specific outcomes related to health, functional status, and quality of life resulting from a patient-centered, intensive care coordination and management intervention correlate with improved linkage to primary care while reducing hospitalizations and emergency department visits. We will then relate these benefits to program costs using standard cost-effectiveness analysis techniques.

Our program model is innovative in its approach, employing Care Management Teams comprised of social workers, community based care managers, and dedicated clinicians who work to meet patients' needs in both the health care setting and the community.

Specific Aim 1

To compare changes in outcomes related to health status, quality of life, and care satisfaction between high-risk intervention patients and controls using quantitative and qualitative methods.

Associated hypotheses Compared to baseline assessments administered at the time of enrollment, 1.1 Intervention patients will have measurable improvements in health status as measured by the SF-12 and the PHQ-9 at 12-month follow-up. Enrollees will have measurable improvements in quality of life as measured by the Perceived Availability of Support scale, the CHAOS scale, and housing status at 12- and 24-month follow-up.

1.2 Intervention patients will have measurable improvements in personal satisfaction with health care as measured by the PSQ-18 at 12 and 24-month follow-up.

Specific Aim 2

To determine if improvements in linkage to primary care (defined as 3 visits to the same clinic within 12 months), and reduced use of acute care services (emergency department visits and hospital admissions) are associated with improved health status, quality of life, and personal satisfaction with health care .

Associated hypotheses 2.1 Improvements in measures of health status are associated with improved linkage to primary care and reductions in use of acute care services.

2.2 Improvements in measures of quality of life are associated with improved linkage to primary care and reductions in use of acute care services.

2.3 Improvements in measures of personal satisfaction are associated with improved linkage to primary care and reductions in use of acute care services.

Specific Aim 3

To understand the economic impact of the intervention by measuring its component financial and societal costs, and to perform a cost- effectiveness analysis for primary and secondary outcomes.

Associated hypotheses 3.1 The overall reduction in health care costs will meet or exceed the cost of the intervention accounting for all intervention-related costs.

3.2 The intervention will have favorable value compared to alternative uses of healthcare resources for this priority population.

3.2.a. The cost of the intervention per hospitalization averted (and associated mortality) will be favorable.

3.2.b The cost of the intervention per improvement in QALY will be favorable

ELIGIBILITY:
Inclusion Criteria:

Fee-for-service Medicaid over age 18 identified as high-risk (risk score over 30 based on validated case-finding algorithm) by the New York State Department of Health, residing in pre-specified zip codes in the HHC catchment area

Exclusion Criteria:

Medicaid enrollees who are not fee-for-service Under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2013-11-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is change in health status as measured by the SF-12. | 6-36 months
  The SF-12 is a shorter yet comparable version of the SF-36 and is an accepted measure for evaluating treatment effectiveness in clinical trials.45-46 The SF-12 has both a mental and physical health component, and provides both a physical component summary (PCS) score and mental component summary (MCS) score. This type of health measure is ideal for this study population, which has high rates of chronic disease including mental health diagnoses.

SECONDARY OUTCOMES:
changes in ED visits and hospitalizations based on Medicaid claims data provided by the New York State Dept of Health | 6-36 months
  We'll evaluate changes in the numbers of ED visits and hospitalizations for enrollees before and after enrollment, and also compare differences between enrollees and those who were eligible for enrollment but not enrolled
changes in primary care outpatient care | 6-36 months
  For intervention enrollees, we'll evaluate changes in the numbers who report they have a primary care provider before and after enrollment, as well as the number of outpatient primary care visits before and after enrollment
self reported health | 6-36 months
  changes in self-reported health using the SF-12 for intervention enrollees comparing the baseline report at time of enrollment to 6-12 month intervals after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Raven, MD, MPH, MSc, Principal Investigator — NYU SOM, HHC, UCSF
Locations (1):
- New York City Health and Hospitals Corporation Central Office, Office of Medical and Professional Affairs, New York, New York, United States

REFERENCES:
- [Background] Raven MC, Billings JC, Goldfrank LR, Manheimer ED, Gourevitch MN. Medicaid patients at high risk for frequent hospital admission: real-time identification and remediable risks. J Urban Health. 2009 Mar;86(2):230-41. doi: 10.1007/s11524-008-9336-1. Epub 2008 Dec 12. PMID 19082899
- [Background] Raven MC, Carrier ER, Lee J, Billings JC, Marr M, Gourevitch MN. Substance use treatment barriers for patients with frequent hospital admissions. J Subst Abuse Treat. 2010 Jan;38(1):22-30. doi: 10.1016/j.jsat.2009.05.009. Epub 2009 Jun 21. PMID 19540700
- [Background] Billings J, Mijanovich T. Improving the management of care for high-cost Medicaid patients. Health Aff (Millwood). 2007 Nov-Dec;26(6):1643-54. doi: 10.1377/hlthaff.26.6.1643. PMID 17978384